CLINICAL TRIAL: NCT01992887
Title: Retention and Engagement in Care of Patients Prior to ART Initiation in the Kagera Region of Tanzania
Brief Title: Pre-ART Retention in Care in Tanzania
Acronym: PARC
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Ministry of Health and Social Welfare, Tanzania (Other Government); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Batya Elul, Assistant Professor of Clinical Epidemiology, Columbia University
Other Study IDs: AAAI0251; 3R01MH089831 (NIH)
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: HIV (Human Immunodeficiency Virus); AIDS (Acquired Immunodeficiency Syndrome)
Keywords: HIV/AIDS; Retention; ART (anti-retroviral therapy) ineligible
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- In-depth Interview: Up to 20 in-depth interviews will be conducted among adult ART naïve patients, balanced by gender, site and reason for ART naiveté (determined ineligible or eligibility not yet determined) as much as possible. Up to 4 in-depth interviews will be conducted with health care providers.
- Focus Group Participants: Up to 40 patients ineligible or not yet eligible for ART will be invited to join a focus group discussion. Patients will be eligible for selection for either in-depth interviews or focus group discussions if they have made at least one prior visit to the clinic. Selected patients will be balanced as much as possible by gender and by pre-ART status (e.g. roughly half pre-ART eligibility determined, and roughly half pre-ART eligibility indeterminate).
- Prospective Cohort: Based on historical patient data from the four study CTCs, we expect that approximately 1,000 patients will enroll in HIV care at these clinics during the study period and be determined not eligible for ART or of unknown eligibility. Assuming a 10% refusal rate, approximately 900 patients would then enroll in this study and complete baseline interviews. These 900 patients will be prospectively monitored using routinely collected patient care data for up to 24 months. Outreach workers will attempt to trace all of the enrolled patients who are observed to be LTF during the study period, and complete a defaulter tracing survey.

SUMMARY:
Retention of patients in HIV care following diagnosis and enrollment is critical to the long-term success of HIV care and treatment scale-up. The goal of this study is to better understand the factors that influence retention and engagement in HIV care among adult patients who are enrolled in HIV care and are not yet eligible for antiretroviral therapy (ART). The study will be conducted at four HIV care and treatment clinics (CTCs) in Kagera Region, Tanzania. This is a mixed-methods study with both qualitative (interviews) and quantitative (surveys) data collection. Our findings will be important towards designing programs that help patients remain in HIV care.

DETAILED DESCRIPTION:
Retention of patients in HIV care following diagnosis and enrollment is a chronic challenge in both resource rich and resource poor settings (Rosen, Fox et al. 2007; WHO 2009; Fox and Rosen 2010), and is critical to the long-term success of HIV care and treatment scale-up. Most research on retention in care has focused on persons who are eligible for or have initiated antiretroviral therapy (ART), generally examined only demographic and clinical determinants. However, a large proportion of patients enrolled in HIV care (e.g., 45%, according to our data from 722 sub-Saharan African clinics) have not been determined to be ART-eligible and have not yet initiated ART; among these individuals, even less is known about the magnitude and determinants of non-retention in care. Retention in HIV care prior to ART initiation is a pre-requisite to: 1) optimal prophylaxis, diagnosis, and treatment of opportunistic illnesses (OIs); 2) effective secondary prevention of HIV transmission, such as by patient counseling and education, earlier diagnosis of infected family members and sexual partners, and prevention of mother to child transmission (PMTCT); and 3) more timely ART initiation. Retention in care among patients at earlier disease stages is also increasingly important given the WHO-recommended expansion of ART eligibility guidelines in resource-limited settings (WHO 2009).

Objective: The goal of this study is to better understand barriers and enablers to retention and engagement in HIV care among adult patients who are enrolled in HIV care and are not yet eligible for ART. The specific objectives are:

1. To describe themes in barriers and enablers to retention and engagement in HIV care;
2. To conduct structured interviews to gather relevant baseline information on potential determinants of non-retention and non-engagement in HIV care;
3. To estimate the incidence of short-term outcomes (missed visits and lost to follow-up (LTF)), including the rate and proportion of those LTF who are no longer engaged in HIV care; and
4. To identify determinants of missed visits, LTF, and non-engagement in care among ART-ineligible patients.

Methods: This study will be conducted using qualitative and quantitative methods at four HIV care and treatment clinics (CTCs) in Kagera Region, Tanzania.

1. Qualitative: in-depth interviews at two CTCs with up to 20 adult patients (ART naïve, and ineligible or indeterminate for ART) and about 4 health care workers; and focus group discussions (about 4 groups of about 6-10 persons/group) with adult patients (ART naïve, and ineligible or indeterminate for ART).
2. Quantitative: 1) structured baseline interviews at four CTCs (n= approximately 900 adult patients who are ART naïve, and ineligible or indeterminate for ART); 2) prospective monitoring of these 900 patients using routine CTC patient data to assess missed visits and LTF; and 4) brief structured surveys of patients who become LTF and are reached through defaulter tracing efforts.

ELIGIBILITY:
QUALITATIVE COHORT

In-depth key informant interviews and focus groups will be conducted with patients that meet the following criteria:

ART-eligibility indeterminate patients (n= approximately 10 in-depth and up to 20 focus group participants, where half are from a rural site, Mugana District Hospital and half are from an urban site, Nyakahanga District Hospital)

i) Inclusion criteria:

* ≥18 years of age
* ART naïve (unless for prior PMTCT)
* made at least one clinic visit prior to study enrollment
* unknown ART eligibility,
* willing to give informed consent.

ii) Exclusion criteria:

* <18 years of age
* initiated ART other than PMTCT prior to enrollment
* have known ART eligibility or ineligibility
* not willing to give informed consent.

ART-ineligible patients (n= approximately 10 in-depth and up to 20 focus group participants, where half are from a rural site, Mugana District Hospital and half are from an urban site, Nyakahanga District Hospital)

i) Inclusion criteria:

* ≥18 years of age
* ART naïve (unless for prior PMTCT)
* made at least one clinic visit prior to study enrollment
* known ART ineligibility
* willing to give informed consent.

ii) Exclusion criteria:

* <18 years of age
* initiated ART other than PMTCT prior to enrollment
* have known ART eligibility
* not willing to give informed consent

Health care workers will be purposefully selected for participation according to the following criteria:

i) Inclusion criteria:

* ≥18 years of age
* have worked at that HIV clinic more than any other post within the hospital for at least 6 months
* medical officer, clinical officer or nurse
* willing to give informed consent.

ii) Exclusion criteria:

* <18 years of age
* primarily posted at another clinic (just part-time or tempory assignment to HIV clinic)
* not willing to give informed consent

PROSPECTIVE COHORT

Patients that meet the following criteria will be included in the prospective study cohort:

i) Inclusion criteria:

* ≥18 years of age
* ART naïve (unless for prior PMTCT)
* enrolled in the study CTC
* ART-ineligible or of indeterminate ART eligibility
* willing to provide written informed consent,contact information and accept a home visit to verify outcomes if they become LTF.

ii) Exclusion criteria:

* <18 years of age
* initiated ART other than PMTCT prior to study enrollment
* ART eligible
* and/ or not willing to provide written informed consent, contact information or accept a home visit if LTF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at four HIV CTCs in the Kagera region of northwestern Tanzania. The 8,000 patients enrolled in HIV care at these clinics represent 30% of HIV patients ever enrolled in ICAP-supported clinics across Kagera Region. Patients will be eligible for selection for either in-depth interviews or focus group discussions if they have made at least one prior visit to the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 948 (Actual)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of those lost to follow-up (LTF) who are no longer engaged in HIV care | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Batya Elul, PhD, MSc, Principal Investigator — ICAP-NY, Columbia University
Locations (4):
- Tanzania (4):
  - Ndolage District Hospital, Kamachumu, Kagera
  - Mugana District Hospital, Mugana, Kagera
  - Nyakahanga District Hospital, Nyakahanga, Kagera
  - Rubya District Hospital, Rubya, Kagera

REFERENCES:
- [Background] Fox MP, Rosen S. Patient retention in antiretroviral therapy programs up to three years on treatment in sub-Saharan Africa, 2007-2009: systematic review. Trop Med Int Health. 2010 Jun;15 Suppl 1(s1):1-15. doi: 10.1111/j.1365-3156.2010.02508.x. PMID 20586956
- [Background] Rosen S, Fox MP, Gill CJ. Patient retention in antiretroviral therapy programs in sub-Saharan Africa: a systematic review. PLoS Med. 2007 Oct 16;4(10):e298. doi: 10.1371/journal.pmed.0040298. PMID 17941716
- [Background] Antiretroviral Therapy for HIV Infection in Adults and Adolescents: Recommendations for a Public Health Approach: 2010 Revision. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138540/ PMID 23741771
- [Background] WHO (2009). Towards Universal Access: Scaling up priority HIV/AIDS Interventions in the Health Sector: Progress report 2009. Geneva, WHO.